CLINICAL TRIAL: NCT04039009
Title: Apical Pelvic Compartment Support in Infertility Patients
Brief Title: Apical Pelvic Support in Infertility Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Adnan Orhan, Principal Investigator. Associate professor, Obstetrician and Gynecologist, Uludag University
Other Study IDs: UU-MREC-2019-9/22
Record Dates: First submitted 2019-07-28; First posted 2019-07-31 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Infertility, Female; Pelvic Organ Prolapse; Pelvic Floor Disorders
Keywords: Pelvic organ prolapse; Infertility; Apical pelvic support
MeSH Terms: conditions — Infertility, Female; Pelvic Organ Prolapse; Pelvic Floor Disorders; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infertility patients: Infertility patients will be examined according to the pelvic organ prolapse quantification classification system during hysteroscopy.
  Interventions: Diagnostic Test: Pelvic Organ Prolapse Quantification system

INTERVENTIONS:
Diagnostic Test: Pelvic Organ Prolapse Quantification system — The Pelvic Organ Prolapse Quantification system assessment tool measures nine anatomical points and distances in the vagina. The hymen is the reference point to which the other points are compared. The prolapsed organs are measured in centimeters to the hymen with an examination ruler.

SUMMARY:
This study aims to evaluate apical pelvic compartment support in infertility patients at the time of hysteroscopy. Apical pelvic compartment evaluation for pelvic organ prolapse will be performed in infertility patients undergoing hysteroscopy.

DETAILED DESCRIPTION:
The incidence of pelvic organ prolapse in the whole population has been demonstrated several times in previous studies. However, pelvic floor defects in young infertility patients are not known. In this study, a clinical pelvic floor assessment with the pelvic organ quantification system will be performed in infertility patients during standard physical examinations or hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-45
* Patients who cannot become pregnant despite regular sexual intercourse for more than one year

Exclusion Criteria:

* Malignity
* Patients who become pregnant during infertility assessment

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Patients examined for female infertility will be included in the study.
Study Population: The study population is the patients examined for female infertility.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Stages of the pelvic organ prolapse | 2 minutes
  Once the measurements are taken, the infertility patients are assigned to the corresponding POP-Q stage. Stage-0 is no prolapse. Stage-1 stands for the most distal portion of the prolapse is more than 1 cm above the level of the hymen. Stage-2 stands for the most distal prolapse is between 1 cm above and 1 cm below the hymen (at least one point is -1, 0, or +1). Stage-3: The most distal prolapse is more than 1 cm below the hymen but no further than 2 cm less than total vaginal length. Stage-4 stands for the complete vaginal eversion.

CONTACTS AND LOCATIONS:
Overall Officials: Gurkan Uncu, Prof., Study Director — ULUDAG UNIVERSITY HOSPITAL BURSA TURKEY
Locations (1):
- Uludag University Hospital, Department of Obstetrics and Gynecology, Bursa, Ozluce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nygaard I, Barber MD, Burgio KL, Kenton K, Meikle S, Schaffer J, Spino C, Whitehead WE, Wu J, Brody DJ; Pelvic Floor Disorders Network. Prevalence of symptomatic pelvic floor disorders in US women. JAMA. 2008 Sep 17;300(11):1311-6. doi: 10.1001/jama.300.11.1311. PMID 18799443
- [Background] Swift SE. The distribution of pelvic organ support in a population of female subjects seen for routine gynecologic health care. Am J Obstet Gynecol. 2000 Aug;183(2):277-85. doi: 10.1067/mob.2000.107583. PMID 10942459